CLINICAL TRIAL: NCT01307345
Title: Remote Monitoring and Contingency Management Reinforcement for Alcohol Abstinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-058-1; P30DA023918 (NIH)
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Alcohol Use
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monitoring Alone (No Intervention): Research assistants will phone or text participants and request videorecordings of breathalyzer samples up to 21 times per week. Participants will receive compensation for each valid videorecording that occurs within the requested one-hour time frame, and bonus compensation each time all requested videorecordings are submitted within the timeframe over a 7-day period, and/or if >90% of prompts are returned over the study period.
- Monitoring plus contingency management for abstinence (Experimental): Participants assigned to this condition will receive the same monitoring schedule outlined above, plus the same payment for compliance. In addition, they will receive contingent reinforcement for submission of videorecordings that demonstrate negative breath alcohol samples. For each sample submitted that reads below the cut point, participants will receive vouchers for payment.
  Interventions: Behavioral: contingency management for abstinence

INTERVENTIONS:
Behavioral: contingency management for abstinence — For each breath sample submitted that reads below the cut point, participants will receive a voucher that can be exchanged for a check or gift card. Amounts earned will increase for each consecutive negative sample submitted, up to a maximum amount.
  Arms: Monitoring plus contingency management for abstinence

SUMMARY:
This pilot project proposes to monitor real-world alcohol use using a novel technology-cell phone videorecordings in conjunction with breathalyzer recordings-and to conduct a small randomized study of this technology for reinforcing alcohol abstinence. Individuals with frequent alcohol use (N = 30) will be asked to carry a study cell phone plus a handheld breathalyzer for one month. Participants will be randomized to one of two conditions: alcohol monitoring or alcohol monitoring plus contingency management. In both conditions, research assistants will telephone participants on their cell phone an average of 10 times per week to request submission of a breathalyzer sample using the video monitoring function on the cell phone. Samples will be time and date stamped, and the video containing the breathalyzer result will be sent to study staff via the cell phone. Participants will be compensated for each video recorded within one hour of receiving the prompt. Participants randomized to the contingency management condition will receive the same alcohol monitoring described above, and they will also receive reinforcement for each alcohol negative breath sample submitted within one hour of the prompt. Data from this pilot project will be useful for (1) determining the feasibility of assessing alcohol use in the natural environment via breathalyzers and cell phone technology, and (2) estimating effect sizes of a CM intervention that reinforces alcohol abstinence using breathalyzers and cell phone technology. In an exploratory manner, we will also evaluate the reliability and validity of the video monitoring procedure and trends toward changes in psychosocial functioning.

ELIGIBILITY:
Inclusion Criteria:

* age >21 years
* frequent alcohol use
* willing to use a cell phone and breathalyzer for 28 days
* have a valid photo ID (driver's license, passport, state ID)
* are willing to sign an off-campus property transfer form and return study equipment in four weeks

Exclusion Criteria:

* desire for, or have received, treatment for alcohol use in the past 6 months
* non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
proportion of negative breath samples submitted | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Alessi, Ph.D., Principal Investigator — University of Conncecticut Health Center
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Derived] Alessi SM, Petry NM. A randomized study of cellphone technology to reinforce alcohol abstinence in the natural environment. Addiction. 2013 May;108(5):900-9. doi: 10.1111/add.12093. Epub 2013 Jan 30. PMID 23279560